CLINICAL TRIAL: NCT03622268
Title: Assessing the Appropriate Energy Expenditure Requirement Using Indirect Calorimetry for Liver Transplant Recipients
Brief Title: Using Indirect Calorimetry for Liver Transplants Patients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, Associate professor, Asan Medical Center
Other Study IDs: AsanMC-LTindirectKcal
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Indirect Calorimetry
Keywords: indirect calorimetry; energy expenditure assessment; intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indirect calorimetry measurement: Using indirect calorimetry for measure resting energy expenditure

SUMMARY:
Although predicted REE calculated using the Penn state 1988 method agreed (ICC 0.61, p=0.00014) with the measured REE, all three predictive equations had a fixed bias and appeared to be inaccurate for predicting REE for liver transplant recipients.

Therefore, precise measurements using indirect calorimetry may be helpful when treating critically ill patients to avoid underestimating or overestimating their metabolic needs.

DETAILED DESCRIPTION:
Rationale: The aim of this study was to compare predictive equations with indirect calorimetry and identify the appropriate energy expenditure requirement of liver transplant(LT) recipients in South Korea.

Methods: This prospective observational study was conducted in a surgical ICU in an academic tertiary hospital over three months. Thirty mechanically ventilated patients who had received liver transplants and were expected to stay in the ICU more than 2 days were studied. Resting energy expenditure(REE) was measured 48 hours after ICU admission using open-circuit indirect calorimetry. Theoretical REE was estimated using three predictive equations: Harris-Benedict methods, lreton-Jones ventilated, and Penn state 1988. The REEs derived from each predictive equation were compared with the measured REE using an intraclass correlation coefficient (ICC) and a Bland-Altman plot.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients who had received liver transplants and were expected to stay in the ICU more than 2 days were studied.

Exclusion Criteria:

* Refusal
* patients who were extubated before 36 hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had received liver transplants
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Comparing REE with the measurement for each predictive equation and indirect calorimetry | 1 year
  The REEs derived from each predictive equation were compared with the measured REE using an intraclass correlation coefficient (ICC) and a Bland-Altman plot.

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyung Hong, Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Hakjae Lee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McClave SA, Martindale RG, Kiraly L. The use of indirect calorimetry in the intensive care unit. Curr Opin Clin Nutr Metab Care. 2013 Mar;16(2):202-8. doi: 10.1097/MCO.0b013e32835dbc54. PMID 23340008
- [Result] Sundstrom M, Tjader I, Rooyackers O, Wernerman J. Indirect calorimetry in mechanically ventilated patients. A systematic comparison of three instruments. Clin Nutr. 2013 Feb;32(1):118-21. doi: 10.1016/j.clnu.2012.06.004. Epub 2012 Jul 3. PMID 22763268
- [Result] Kross EK, Sena M, Schmidt K, Stapleton RD. A comparison of predictive equations of energy expenditure and measured energy expenditure in critically ill patients. J Crit Care. 2012 Jun;27(3):321.e5-12. doi: 10.1016/j.jcrc.2011.07.084. Epub 2012 Mar 14. PMID 22425340
- [Result] Xiao GZ, Su L, Duan PK, Wang QX, Huang Y. [Comparison of measuring energy expenditure with indirect calorimetry and traditional estimation of energy expenditure in patients in intensive care unit]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2011 Jul;23(7):392-5. Chinese. PMID 21787465